CLINICAL TRIAL: NCT06697119
Title: Efficacy and Safety of Fecal Microbiota Transplantation in Patients with Irritable Bowel Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-2210-784-004
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Disease
Keywords: fecal microbiota transplantation; FMT; IBS; Irritable bowel disease
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT (Experimental): Fecal microbiota transplantation: fecal suspension delivered to duodenal 3rd portion via esophagogastroduodenoscopy
  Interventions: Other: Fecal Microbial Transplantation

INTERVENTIONS:
Other: Fecal Microbial Transplantation — Fecal suspension is delivered to duodenal 3rd portion via esophagogastroduodenoscopy

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of fecal microbiota transplantation (FMT) for patients with irritable bowel syndrome (IBS). The main objectives of the study are:

To determine if FMT can significantly reduce IBS symptoms and improve patients' quality of life.

To evaluate any potential adverse effects associated with FMT in IBS patients. Researchers will compare outcomes in patients receiving FMT with a standard care protocol to gauge the effectiveness of FMT in alleviating IBS symptoms.

Participants will:

Receive FMT via endoscopic methods as per the study protocol. Attend scheduled clinic visits for assessments and symptom tracking over a 48-week period, with optional long-term follow-up for up to 3 years.

Complete regular questionnaires and microbiota assessments to monitor symptoms and gut health changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Korean men and women aged 19 to 80 years
2. Diagnosed according to Rome IV criteria, with abdominal pain occurring at least once per week that began more than 6 months prior and has recurred over the past 3 months, accompanied by at least two of the following symptoms: pain related to defecation, changes in stool frequency (increase or decrease), or changes in stool form (looser or harder consistency)
3. Patients with moderate to severe IBS (IBS-SSS score of 175 or higher) with diarrhea-predominant, mixed-type, or abdominal bloating as the main symptom, who have not responded to IBS medication therapy for over 3 months
4. Patients who have had a colonoscopy within the past 5 years, or those who will undergo a colonoscopy after joining the study, and for whom no structural abnormalities in the colon are identified (records from other hospitals within the past 5 years may be used). *Patients who have undergone a biopsy or polypectomy during colonoscopy and can provide examination results are eligible if deemed appropriate by the clinician
5. Females who are surgically infertile or females of childbearing potential with a negative pregnancy test (urine hCG or serum b-hCG); females of childbearing potential or males who agree to use effective contraception (e.g., oral contraceptives, IUD, double-barrier methods, or hormonal implants) during the study period
6. Individuals capable of clearly expressing their intentions without significant neurological or psychiatric issues. Those with neurological or psychiatric conditions may participate if deemed stable with appropriate medication or other treatments
7. Patients who voluntarily provide written informed consent to participate in the study

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Patients who have received investigational drugs within 3 months prior to Visit 1 (if investigational drugs were used within 3 months, consult the study monitor for case-by-case assessment)
3. Patients whom the investigator deems to be at risk or to have conditions that would interfere with participation in the clinical trial
4. Patients with severe congestive heart failure or severe angina
5. Patients diagnosed with lactose intolerance or those who are immunocompromised
6. Patients currently taking medications that may affect the study drug (e.g., intestinal drugs, probiotics), or those who need to continue these medications during the study period. Patients who are currently on these medications can participate after a 2-week washout period
7. Patients whose systolic blood pressure exceeds 160 mmHg or diastolic blood pressure exceeds 100 mmHg at Visit 1, with uncontrolled hypertension regardless of treatment status
8. Patients with uncontrolled endocrine disorders (e.g., diabetes), metabolic disorders (e.g., secondary hyperlipidemia), or hypothyroidism. Patients with a history of hypothyroidism may participate if they have been on a stable thyroid hormone replacement therapy for at least 4 weeks before Visit 2 and have a TSH level within the normal range at Visit 2
9. Patients with impaired renal function (creatinine > 2.0 mg/dL) or nephrotic syndrome at Visit 1
10. Patients with a history of cancer within the last 5 years (except for those deemed cured)
11. Patients with significant psychiatric instability or psychiatric disorders not adequately controlled with medication or other treatment
12. Patients who have taken systemic steroid medications within 1 month prior to Visit 1
13. Patients who have undergone abdominal surgery other than appendectomy, cholecystectomy, cesarean section, hernia repair, or hysterectomy. *Patients with other abdominal surgeries may still participate if deemed eligible by the investigator
14. Any other patient whom the investigator deems unsuitable for the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Changes of IBS-SSS | 12weeks after FMT
  At 12 weeks post-FMT, overall satisfaction with the improvement in IBS symptoms will be evaluated, alongside changes in the IBS Symptom Severity Score (IBS-SSS) to comprehensively assess the effects of FMT on individual IBS symptoms.

SECONDARY OUTCOMES:
Change in IBS-SSS | 4 weeks, 24 weeks, 48 weeks, 2 years, and 3 years after FMT
  Change in IBS-SSS Score for IBS Patients (evaluated by the IBS-SSS questionnaire)
Changes in Stool Frequency and Form | 4 weeks, 12 weeks, 24 weeks, 48 weeks, 2 years, and 3 years after FMT
  Changes in Stool Frequency and Form for IBS Patients (evaluated by the BSFS questionnaire)
Changes in Quality of Life | 4 weeks, 12 weeks, 24 weeks, 48 weeks, 2 years, and 3 years after FMT
  Changes in Quality of Life for IBS Patients (evaluated by the IBS-QoL questionnaire)
Changes in Anxiety and Derpession | 4 weeks, 12 weeks, 24 weeks, 48 weeks, 2 years, and 3 years after FMT
  Changes in Mental Health for IBS Patients (evaluated by the HADS questionnaire)
Changes in gut microbiota | at baseline, 4 weeks, and 12 weeks after FMT
  Differences in Gut Microbiota Between Responders and Non-Responders

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu J, Lv L, Wang C. Efficacy of Fecal Microbiota Transplantation in Irritable Bowel Syndrome: A Meta-Analysis of Randomized Controlled Trials. Front Cell Infect Microbiol. 2022 Feb 28;12:827395. doi: 10.3389/fcimb.2022.827395. eCollection 2022. PMID 35295757
- [Background] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769
- [Background] Aroniadis OC, Brandt LJ, Oneto C, Feuerstadt P, Sherman A, Wolkoff AW, Kassam Z, Sadovsky RG, Elliott RJ, Budree S, Kim M, Keller MJ. Faecal microbiota transplantation for diarrhoea-predominant irritable bowel syndrome: a double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):675-685. doi: 10.1016/S2468-1253(19)30198-0. Epub 2019 Jul 17. PMID 31326345
- [Background] Halkjaer SI, Christensen AH, Lo BZS, Browne PD, Gunther S, Hansen LH, Petersen AM. Faecal microbiota transplantation alters gut microbiota in patients with irritable bowel syndrome: results from a randomised, double-blind placebo-controlled study. Gut. 2018 Dec;67(12):2107-2115. doi: 10.1136/gutjnl-2018-316434. Epub 2018 Jul 6. PMID 29980607
- [Background] Holvoet T, Joossens M, Vazquez-Castellanos JF, Christiaens E, Heyerick L, Boelens J, Verhasselt B, van Vlierberghe H, De Vos M, Raes J, De Looze D. Fecal Microbiota Transplantation Reduces Symptoms in Some Patients With Irritable Bowel Syndrome With Predominant Abdominal Bloating: Short- and Long-term Results From a Placebo-Controlled Randomized Trial. Gastroenterology. 2021 Jan;160(1):145-157.e8. doi: 10.1053/j.gastro.2020.07.013. Epub 2020 Jul 15. PMID 32681922